CLINICAL TRIAL: NCT04827108
Title: Psychometric Properties of the Chinese Version of the Pediatric Nausea Assessment Tool (PeNAT) to Measure Nausea and Vomiting in Hong Kong Chinese Children Undergoing Chemotherapy
Brief Title: Psychometric Properties of the Chinese Version of PeNAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Research Assistant Professor, The Hong Kong Polytechnic University
Other Study IDs: PeNAT validation
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Child; Nausea; Vomiting
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PeNAT validation — Children will be required to fill in a set of questionnaires including the Chinese version of the Pediatric Nausea Assessment Tool (PeNAT), the Chinese version of the Pediatric Quality of Life Inventory 4.0 Cancer Module (PedsQL 4.0), and the Chinese version of Center for Epidemiological Studies Depression Scale for Children (CES-DC)

SUMMARY:
Cancer is a leading cause of death for children. Chemotherapy is the most common treatment for cancer. Notwithstanding the improved survival, children with cancer still have to face a significant amount of symptoms associated with chemotherapy. Two major symptoms induced by chemotherapy are nausea and vomiting. These two symptoms were demonstrated to cause serious disruption in patients' daily function and quality of life. Given these devastating impacts, intervening children with appropriate methods to alleviate nausea and vomiting during chemotherapy is therefore crucial. It is imperative for nurses to develop non-pharmacological interventions to reduce nausea and vomiting, with the goal of improving the QoL of children with cancer when undergoing chemotherapy First, however, careful assessment of nausea and vomiting in children with cancer is a necessary step towards designing appropriate interventions. This study aims to translate and validate an instrument (PeNAT) which can assess nausea and vomiting among Hong Kong Chinese children and adolescents undergoing chemotherapy

DETAILED DESCRIPTION:
Currently, the most effective anti-emetics appear to be 5-HT3 inhibitors, followed by NK1 inhibitors and neuroleptic drugs. Nevertheless, anti-emetics alone are not sufficient to manage these two symptoms. This poor symptom control could be due to healthcare professionals' perception that nausea and vomiting are solely biological problems, and their heavy reliance on pharmacological treatment for management. After literature search, we can identify only one validated instrument, the Pediatric Nausea Assessment tool (PeNAT), assessing chemotherapy-induced nausea and vomiting in children. Yet, this instruments is not available in Chinese. This study aims to translate and validate an instrument (PeNAT) which can assess nausea and vomiting among Hong Kong Chinese children and adolescents undergoing chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Aged 4 - 17
* A confirmed diagnosis of cancer
* Currently undergoing chemotherapy
* Able to speak Cantonese and read Chinese

Exclusion Criteria:

* Cognitive or behavioral problems in medical records

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study targets to recruit 150 subjects from the Hong Kong Children's Hospital.
  Children who meet the inclusion criteria will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
The Chinese version of the Pediatric Nausea Assessment Tool (PeNAT) at baseline | at baseline
  Children will be required to fill in the Chinese version of the Pediatric Nausea Assessment Tool (PeNAT) at baseline. The score ranges from 1 to 4. Higher scores represent a more severe nausea.

SECONDARY OUTCOMES:
The Chinese version of the Pediatric Quality of Life Inventory 4.0 Cancer Module (PedsQL 4.0) at baseline | at baseline
  Children will be required to fill in the Chinese version of Pediatric Quality of Life Inventory 4.0 Cancer Module (PedsQL 4.0) at baseline. The score ranges from 0 to 100. Higher scores represent a better quality of life.
The Chinese version of Center for Epidemiological Studies Depression Scale for Children (CES-DC) at baseline | at baseline
  Children will be required to fill in the Chinese version of Center for Epidemiological Studies Depression Scale for Children (CES-DC) at baseline. The score ranges from 0 to 60. Higher scores represent a higher number of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Lam, PhD, Principal Investigator — The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No